CLINICAL TRIAL: NCT02233153
Title: Elder-friendly Approaches to the Surgical Environment - Implementation of an Elder Friendly Surgical Unit
Brief Title: Elder-friendly Approaches to the Surgical Environment (EASE) Study
Acronym: EASE
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Rachel Khadaroo, Assistant Professor, University of Alberta
Other Study IDs: Pro00047180
Record Dates: First submitted 2014-08-22; First posted 2014-09-08 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: General Surgery
Keywords: Senior; Elderly; Acute Care; Emergency Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-Elder Friendly Surgical Intervention Group: Elder Acute Care and Emergency Surgery patients
- Post-Elder Friendly Surgical Intervention Group: Elder Acute Care and Emergency Surgery patients
  Interventions: Other: Elder-Friendly Surgical Unit
- Pre-Elder Friendly Surgical Control Group: Elder Acute Care and Emergency Surgery patients
- Post-Elder Friendly Surgical Control Group

INTERVENTIONS:
Other: Elder-Friendly Surgical Unit
  Groups: Post-Elder Friendly Surgical Intervention Group

SUMMARY:
The aim of this study is to examine the impact implementing an elder-friendly surgical unit has on post-operative complications, mortality and quality of life for patients ≥ 65 years old who have undergone emergency surgical care.

DETAILED DESCRIPTION:
The investigators hypothesize that the elder-friendly surgical unit will reduce in-hospital complications and mortality in a cost-effective manner, for this at risk population.

Specific elder-friendly interventions include:

1. Locate all elderly surgical patients on one nursing unit
2. Interdisciplinary team-based care
3. Elder-friendly evidence-informed practices including: comfort rounds with early mobilization, delirium prevention/management, optimal nutrition and prevention of post-operative complications
4. Early and interdisciplinary discharge management

This is a prospective, before-after study with a concurrent control group. Four senior patient groups will be followed:

ELIGIBILITY:
Inclusion Criteria:

* All patients > 65 years old admitted for Acute care and Emergency Surgery
* Received acute abdominal surgery

Exclusion Criteria:

* Elective general surgery cases
* Nursing home resident requiring full nursing care [dependency in 3 or more activities of daily living ]
* Palliative surgery [surgery with the primary intention of improving quality of life or relieving symptoms caused by advancing non-curative disease]
* Multi-system trauma
* Patients from out of province or transferred from another inpatient service or hospital

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients > 65 years old admitted and received acute abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 723 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Post-Operative complications | During initial in-hospital stay (0-12 weeks on average)
  Includes a) intensive care unit admission (includes respiratory failure, cardiac arrest or septic shock), b) vascular complications (myocardial infarction, stroke, deep venous thrombosis, pulmonary embolism), c) serious infections (pneumonia, intra-abdominal abscess, urinary tract infection, deep wound infection or infected decubitus ulcer) or d) protracted delirium (≥48 hours)
Death | During initial in-hospital stay (0-12 weeks on average)

SECONDARY OUTCOMES:
Post-discharge complications or health-events requiring re-admission | Within 30 days post-discharge
Cost per quality-adjusted life year | 6 months post-discharge
  Both direct and indirect study participant costs

OTHER OUTCOMES:
Health Related Quality of Life | 6 weeks and 6 months post-discharge
  Including: EQ-5D questionnaire, SF-12 Questionnaire
Functional Status (Frailty) | 6 weeks post-discharge
  Including: Edmonton Frail Scale, and Timed Up-and-Go Test

CONTACTS AND LOCATIONS:
Overall Officials: Rachel G Khadaroo, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Foothills Medical Center, Acute Care Emergency Surgical Services, Calgary, Alberta
  - University of Alberta Hospital, Acute Care and Emergency Surgery Service, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanson HM, Warkentin L, Wilson R, Sandhu N, Slaughter SE, Khadaroo RG. Facilitators and barriers of change toward an elder-friendly surgical environment: perspectives of clinician stakeholder groups. BMC Health Serv Res. 2017 Aug 24;17(1):596. doi: 10.1186/s12913-017-2481-z. PMID 28836979
- [Background] Khadaroo RG, Padwal RS, Wagg AS, Clement F, Warkentin LM, Holroyd-Leduc J. Optimizing senior's surgical care - Elder-friendly Approaches to the Surgical Environment (EASE) study: rationale and objectives. BMC Health Serv Res. 2015 Aug 21;15:338. doi: 10.1186/s12913-015-1001-2. PMID 26293153
- [Result] Li Y, Pederson JL, Churchill TA, Wagg AS, Holroyd-Leduc JM, Alagiakrishnan K, Padwal RS, Khadaroo RG. Impact of frailty on outcomes after discharge in older surgical patients: a prospective cohort study. CMAJ. 2018 Feb 20;190(7):E184-E190. doi: 10.1503/cmaj.161403. PMID 29565018
- [Result] Eamer GJ, Clement F, Pederson JL, Churchill TA, Khadaroo RG. Analysis of postdischarge costs following emergent general surgery in elderly patients. Can J Surg. 2018 Feb;61(1):19-27. doi: 10.1503/cjs.002617. Epub 2017 Dec 1. PMID 29368673
- [Result] McComb A, Warkentin LM, McNeely ML, Khadaroo RG. Development of a reconditioning program for elderly abdominal surgery patients: the Elder-friendly Approaches to the Surgical Environment-BEdside reconditioning for Functional ImprovemenTs (EASE-BE FIT) pilot study. World J Emerg Surg. 2018 May 21;13:21. doi: 10.1186/s13017-018-0180-7. eCollection 2018. PMID 29942346
- [Derived] Pederson JL, Padwal RS, Warkentin LM, Holroyd-Leduc JM, Wagg A, Khadaroo RG. The impact of delayed mobilization on post-discharge outcomes after emergency abdominal surgery: A prospective cohort study in older patients. PLoS One. 2020 Nov 6;15(11):e0241554. doi: 10.1371/journal.pone.0241554. eCollection 2020. PMID 33156849
- [Derived] Khadaroo RG, Warkentin LM, Wagg AS, Padwal RS, Clement F, Wang X, Buie WD, Holroyd-Leduc J. Clinical Effectiveness of the Elder-Friendly Approaches to the Surgical Environment Initiative in Emergency General Surgery. JAMA Surg. 2020 Apr 1;155(4):e196021. doi: 10.1001/jamasurg.2019.6021. Epub 2020 Apr 15. PMID 32049271
- [Derived] Eamer GJ, Clement F, Holroyd-Leduc J, Wagg A, Padwal R, Khadaroo RG. Frailty predicts increased costs in emergent general surgery patients: A prospective cohort cost analysis. Surgery. 2019 Jul;166(1):82-87. doi: 10.1016/j.surg.2019.01.033. Epub 2019 Apr 27. PMID 31036332